CLINICAL TRIAL: NCT00832650
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Multiple Dose Study To Investigate The Effects Of 8 Mg Fesoterodine SR Tablets And 10 Mg Solifenacin Tablet On Gastrointestinal Transit In Healthy Female Subjects.
Brief Title: Multiple Dose Study To Investigate The Effects Of Fesoterodine And Solifenacin On Gastrointestinal Transit
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol A0221057 was terminated on December 25, 2009 for futility. There were no safety concerns related to this decision.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0221057; NCT00892034 (obsolete NCT alias)
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Healthy; Fesoterodine; Solifenacin
MeSH Terms: interventions — fesoterodine; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fesoterodine (Experimental): Tablets
  Interventions: Drug: fesoterodine fumarate
- Placebo (Placebo Comparator): Tablets
  Interventions: Drug: placebo
- Solifenacin (Active Comparator): Tablets
  Interventions: Drug: solifenacin

INTERVENTIONS:
Drug: fesoterodine fumarate — 8 mg OD for 14 days
  Arms: Fesoterodine
Drug: placebo — OD for 14 days
  Arms: Placebo
Drug: solifenacin — 10 mg OD for 14 days
  Arms: Solifenacin

SUMMARY:
To assess the effect of fesoterodine 8 mg as compared to solifenacin 10 mg on colonic transit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects

Exclusion Criteria:

* Evidence or history of clinically significant findings at screening

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Bharucha AE, Isowa H, Hiro S, Guan Z. Differential effects of selective and non-selective muscarinic antagonists on gastrointestinal transit and bowel function in healthy women. Neurogastroenterol Motil. 2013 Jan;25(1):e35-43. doi: 10.1111/nmo.12043. Epub 2012 Nov 21. PMID 23171069
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221057&StudyName=Multiple%20Dose%20Study%20To%20Investigate%20The%20Effects%20Of%20Fesoterodine%20And%20Solifenacin%20On%20Gastrointestinal%20Transit

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine: Fesoterodine 8 mg tablet once daily
- Placebo: Matched placebo tablet or capsule
- Solifenacin: Solifenacin 10 mg capsule once daily
Period: Overall Study
Arm/Group | Fesoterodine | Placebo | Solifenacin
Started | 25 | 12 | 23
Treated | 25 | 12 | 22
Completed | 25 | 12 | 22
Not Completed | 0 | 0 | 1
Not completed — Randomized but not treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fesoterodine | Placebo | Solifenacin | Total
Number analyzed (Participants) | 25 | 12 | 23 | 60
Age, Customized [Number; unit: participants]
  less than 18 years | 0 | 0 | 0 | 0
  18 to 25 years | 5 | 5 | 6 | 16
  26 to 35 years | 7 | 2 | 6 | 15
  36 to 45 years | 7 | 2 | 8 | 17
  greater than 45 years | 6 | 3 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 23 | 60
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Colonic Transit at 24 Hours
Description: Colonic transit: Geometric centre at 24 hours (GC24) was estimated using geometric mean of counts in ascending (AC), transverse (TC), descending (DC) and rectosigmoid (RS) colon and stool (weighted by factors of 1 to 5 respectively). To calculate the geometric centre, the proportion of colonic counts in each colonic region was multiplied by its weighing factor: (% AC *1 + % TC *2 + % DC *3 + % RS *4 + % stool * 5 ) divided by 100.
Time Frame: Day 13 (Day 12 24 hours post-meal)
Population: Intent to treat (ITT) included all randomized subjects. Imputation by overall mean for missing data.
Measure: Mean (Standard Deviation); unit: counts
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 23
counts | 1.98 (0.770) | 2.51 (1.078) | 1.91 (0.515)
Statistical Analysis 1: Comparison: Fesoterodine vs Solifenacin; Null H10: μF8mg=μS10mg where μF8mg and μS10mg are means of GC24 for fesoterodine 8mg and solifenacin 10mg, respectively; Test type: Superiority or Other; ANCOVA; LS Mean difference = 0.051, 95% CI 2-sided [-0.334 to 0.436] — Least squares mean was calculated based on the ANCOVA model with treatment group as a fixed effect and baseline values, age and Body Mass Index (BMI) as covariates

2. Secondary Outcome: Proximal Colonic Emptying Time
Description: Estimated by power exponential analysis of the proportionate emptying over time of counts from the colon.
Time Frame: Day 12 to 14
Population: ITT included all randomized subjects. Imputation by overall mean for missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 23
hours | 21.06 (5.500) | 14.79 (6.239) | 19.23 (6.194)

3. Secondary Outcome: Colonic Transit at 48 Hours
Description: Colonic transit: Geometric centre at 48 hours (GC48) was estimated using geometric mean of counts in ascending (AC), transverse (TC), descending (DC) and rectosigmoid (RS) colon and stool (weighted by factors of 1 to 5 respectively). To calculate the geometric centre, the proportion of colonic counts in each colonic region was multiplied by its weighing factor: (% AC *1 + % TC *2 + % DC *3 + % RS *4 + % stool * 5 ) divided by 100.
Time Frame: Day 14 (Day 12 48 hours post-meal)
Population: ITT included all randomized subjects. Imputation by overall mean for missing data.
Measure: Mean (Standard Deviation); unit: counts
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 23
counts | 3.55 (0.934) | 3.67 (1.066) | 3.14 (0.765)

4. Secondary Outcome: Colonic Filling at 6 Hours
Description: A surrogate marker of small bowel transit time.
Time Frame: Day 12
Population: ITT included all randomized subjects. Imputation by overall mean for missing data.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 23
percentage | 7.84 (16.286) | 69.58 (25.854) | 24.06 (23.696)

5. Secondary Outcome: Time to Gastric Emptying
Description: Ascending colon emptying t½ was estimated by power exponential analysis of the proportionate emptying over time of counts from the colon.
Time Frame: Day 12: 2 hours, 4 hours
Population: ITT included all randomized subjects. Imputation by overall mean for missing data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 23
minutes | 145.00 (32.628) | 112.92 (21.998) | 127.47 (35.456)

6. Secondary Outcome: Mean Number of Stools Per Day
Description: Number of stools passed on each notional day where each visit to the toilet counts as one stool (only) unless nothing is passed. Mean of 3 days.
Time Frame: Day 11 to 13
Population: ITT, all randomized subjects with analyzeable data. Imputation by individual mean for missing data if at least one observation was observed in last 3 days.
Measure: Mean (Standard Deviation); unit: stools
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 22
stools | 0.93 (0.397) | 1.06 (0.422) | 1.11 (0.497)

7. Secondary Outcome: Mean Score of Stool Consistency Per Day
Description: Calculated by averaging the values of the stool form given at each visit to the toilet on each notional day. Mean of 3 days. Range of possible scores: 1 (hard lumps) to 7 (watery).
Time Frame: Day 11 to 13
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 22
score on a scale | 3.66 (1.149) | 3.29 (1.112) | 3.02 (1.057)

8. Secondary Outcome: Average Score of Ease of Passage During Defecation Per Day
Description: Calculated by averaging the values given for the ease of passage at each visit to the toilet on each notional day. Mean of 3 days. Range of possible scores: 1 (Manual disimpaction) to 7 (Incontinent).
Time Frame: Day 11 to 13
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 22
score on a scale | 3.90 (0.403) | 3.97 (0.096) | 3.83 (0.705)

9. Secondary Outcome: Mean Proportion of Bowel Movements With Satisfaction Per Day
Description: The number of stools with satisfaction of "Yes" divided by the total number of stools passed on each notional day. Mean of 3 days.
Time Frame: Day 11 to 13
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mean proportion
Arm/Group | Fesoterodine | Placebo | Solifenacin
Number analyzed (Participants) | 25 | 12 | 22
mean proportion | 0.88 (0.250) | 0.81 (0.324) | 0.93 (0.234)

ADVERSE EVENTS:
Time Frame: Up to 7 days after last dose of study drug
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine | Placebo | Solifenacin
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/12 | 0/22
Other Adverse Events (participants affected / at risk) | 22/25 | 6/12 | 15/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine (N=25) | Placebo (N=12) | Solifenacin (N=22)
Dry eye (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 13 | 0 | 7
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 12 | 3 | 2
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 1 | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated due to futility based on interim analysis with 60 subjects. Although the results of statistical test for the primary endpoint was interpreted, the other endpoint results were interpreted based on statistical inference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.